CLINICAL TRIAL: NCT04375644
Title: Impact of the COVID-19 Pandemic on the Quality of Psychological Life of Healthcare Professionals
Brief Title: Impact of the COVID-19 Pandemic on the Quality of Psychological Life (COVID-PRO-IMPACT)
Acronym: COVIDPROIMPACT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0413
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Covid 19; Stress, Psychological
MeSH Terms: conditions — COVID-19; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires on psychological quality of life — Assessement of evolution of the psychological quality of life of health professionals during the confinement period linked to the COVID-19 pandemic by two questionnaires (one during the confinement period and the second one month after the end of the confinement period)

SUMMARY:
The COVID-19 pandemic is profoundly changing the way people live and work. After the health impact, it is the mental and psychological impact that reaches varying degrees in the entire world population. The previous Asian epidemics have had a lasting impact on the health professionals concerned.

In France, no study has yet assessed the psychological impact of this health crisis on the level of health professionals. Investigators propose to study prospectively the evolution of the state of stress and anxiety of all the professionals practicing within the gynecology-obstetrics departments of 18 French hospitals.

Investigators also hypothesize that the mental repercussions in terms of stress and anxiety within the same service could be different depending on the professional status and the place of exercise (the French regions being impacted in different ways).

In addition to the epidemiological interest, the results of this study may help us to target regions and professionals who will need psychological support during and after this serious health crisis.

ELIGIBILITY:
Inclusion Criteria:

* person over 18
* person exercising a profession in the health field
* person having expressed his non-opposition

Exclusion Criteria:

* inability to understand the information given and the questionnaire
* person deprived of liberty, person under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Person over 18 years of age practicing a health profession in the participating gynecology and obstetrics departments
Sampling Method: Non-Probability Sample
Enrollment: 1565 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Stress state score, during the confinement period | About 10 minutes ( Questionnaire filling time)
  Stress state score, during the confinement period, established by a comparison VAS (visual analogue scale) compared to a period outside COVID-19 (from -5: considerable degradation to +5: considerable improvement, with 0: no change)

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - Gynécologie-Obstétrique CHU de Angers, Angers
  - Gynécologie-Obstétrique Hôpital Pellegrin, Bordeaux
  - Gynécologie-Obstétrique CHRU de Brest, Brest
  - Gynaecology Department, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - Gynécologie-Obstétrique Hôpital Antoine Béclère (APHP), Clamart
  - Gynécologie-Obstétrique CHU Grenoble-Alpes, Hôpital Couple Enfant, La Tronche
  - Gynécologie-Obstétrique Hôpital BICETRE (APHP), Le Kremlin-Bicêtre
  - Gynécologie-Obstétrique Hôpital Jeanne de Flandre - CHRU Lille, Lille
  - Gynécologie-Obstétrique Hôpital de la Mère et de l'Enfant, Limoges
  - Gynécologie-Obstétrique Hôpital de la Croix Rousse, Lyon
  - Gynécologie-Obstétrique Hôpital La Conception, Marseille
  - Gynécologie-Obstétrique Hôpital de la Pitié Salpêtrière (APHP), Paris
  - Gynécologie-Obstétrique Maternité Port-Royal, Groupe Hospitalier Cochin-Broca- Hotel Dieu (APHP), Paris
  - Gynécologie-Obstétrique CHU de Poitiers, Poitiers
  - Gynécologie-Obstétrique CHU Reims - Institut Mère Enfant Alix de Champagne, Reims
  - Gynécologie-Obstétrique CHU de Rennes, Rennes
  - Gynécologie-Obstétrique CHU de Saint Etienne, Saint-Etienne
  - Gynécologie-Obstétrique Hôpital de Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chene G, Nohuz E, Cerruto E, Moret S, Atallah A, Saoud M; French Covid-Pro-Impact Consortium. Psychological impact on healthcare workers in obstetrics and gynecology in France in 18 French University Hospitals during the first Covid-19 lockdown: a prospective observational study. J Psychosom Obstet Gynaecol. 2022 Dec;43(4):433-440. doi: 10.1080/0167482X.2021.2014812. Epub 2021 Dec 16. PMID 34915826